CLINICAL TRIAL: NCT01088945
Title: Safe Passages: Ensuring Quality Transitions From NICU to Ambulatory Care
Brief Title: Safe Passages: Ensuring Quality Transitions From NICU (Neonatal Intensive Care Unit) to Ambulatory Care
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Virginia Moyer (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Virginia Moyer, Professor of Pediatrics (Adjunct), Baylor College of Medicine
Organization: Baylor College of Medicine (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H-26059
Record Dates: First submitted 2010-03-10; First posted 2010-03-18 (Estimated); Last update posted 2015-07-27 (Estimated); Status verified 2015-07

CONDITIONS: Infant, Premature, Diseases
Keywords: Infant, Premature, Diseases
MeSH Terms: conditions — Infant, Premature, Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Enhanced Discharge Process (Experimental): Caregivers of these infants will receive individual coaching in order to enhance their understanding of their infant's problems and enhance their knowledge and skills to care for their fragile infants.
  Interventions: Behavioral: Enhanced Discharge process
- Standard Discharge Process (Active Comparator): These infants will receive the hospital's current standard of care for the discharge of fragile infants from the NICU.
  Interventions: Behavioral: Enhanced Discharge process

INTERVENTIONS:
Behavioral: Enhanced Discharge process — Health Coaching prior to discharge, with an enhanced discharge binder to reinforce the teaching of the Health Coach

SUMMARY:
Infants born prematurely or with complex congenital abnormalities are surviving to discharge in growing numbers and often require significant monitoring and coordination of care in the ambulatory setting. The specific aims of this project are to determine the effectiveness of a redesigned discharge process that includes a Health Coach and an expanded discharge binder to improve health outcomes in the post discharge follow-up period as compared with usual care. The outcomes to be evaluated include the occurrence of adverse events in the post-discharge period, quality of follow up care, and caregiver satisfaction with the process.

DETAILED DESCRIPTION:
Infants born prematurely or with complex congenital abnormalities are surviving to discharge in growing numbers and often require significant monitoring and coordination of care in the ambulatory setting. These complicated infants have spent all of their lives in the hospital setting, and are strangers in their own homes. Although the transition of the fragile child from intensive care specialist to the ambulatory care provider begins at hospital discharge, it is incomplete until the child receives appropriate outpatient follow-up with a primary care pediatrician. Over this prolonged time period, the child is especially vulnerable to errors related to breakdowns in care coordination and communication because the responsibility for the patient's care is often not clearly specified. Our team of investigators has recently completed a Health Care Failure Modes and Effects Analysis (HFMEA) of the transition from neonatal intensive care to the ambulatory environment. We will expand upon the Care Transitions Intervention developed by Coleman et al that addressed the problems of older adults who were discharged from hospital to home. In this model, advanced practice nurses, trained as coaches, taught patients and families to coordinate care for themselves, fostering independence. We will include the use of a personal health record, to include specific instructions to recognize and self-manage the most common problems in this population and we will use information technology (IT) to enhance communication with families and with community providers, in particular the primary care provider. Having identified that lack of knowledge and skills on the part of community providers about how to manage these infants as an important risk point, we will add to the Coleman intervention by providing "just-in-time" information to the primary care providers to enhance their knowledge and skill in managing the common problems of neonatal nursery graduates, provided electronically via the Texas Children's Hospital (TCH) clinical decision support program.

ELIGIBILITY:
Inclusion Criteria:

* Infant hospitalized since birth
* Anticipated total length of stay at least 2 weeks
* Speaks English or Spanish
* Planned follow up physician within the hospital's system

Exclusion Criteria

* follow up physician outside of hospital system
* child in protective custody
* child not anticipated to survive

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 229 (Actual)
Dates: Start 2010-03; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
adverse outcomes in first 30 days after discharge from NICU | 30 days
  unplanned ER visits, Unplanned readmissions, deaths, missed appointments

SECONDARY OUTCOMES:
adherence to recommended practices for care of the fragile newborn | 6 months
  adherence by primary care physicians to recommended practices for management of the fragile NICU graduate
Caregiver assessment of the discharge process | 2-3 and 30 days after discharge
  Using a validated measure, the CTM-Neo, caregivers will be interviewed both shortly after discharge and at 30 days to determine satisfaction with the transition from hospital to home.

CONTACTS AND LOCATIONS:
Overall Officials: Virginia A Moyer, MD, MPH, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States

REFERENCES:
- [Derived] Moyer VA, Papile LA, Eichenwald E, Giardino AP, Khan MM, Singh H. An intervention to improve transitions from NICU to ambulatory care: quasi-experimental study. BMJ Qual Saf. 2014 Dec;23(12):e3. doi: 10.1136/bmjqs-2012-001726. PMID 23832926